CLINICAL TRIAL: NCT04818398
Title: Single-Ascending Dose Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of DS-6016a After Subcutaneous Injection in Healthy Japanese Subjects
Brief Title: Study of Single-Ascending Doses of DS-6016a in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DS6016-A-J101; jRCT2051200155 (Other: Japan Registry of Clinical Trial)
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Fibrodysplasia Ossificans Progressiva; Bone Morphogenetic Protein; Activin Receptor-like Kinase-2
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- DS-6016a dose level 1 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- DS-6016a dose level 2 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- DS-6016a dose level 3 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- DS-6016a dose level 4 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- DS-6016a dose level 5 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- DS-6016a dose level 6 (Experimental): Participants will be randomized to receive a single, subcutaneous injection of DS-6016a.
  Interventions: Drug: DS-6016a
- Placebo (Placebo Comparator): Participants will be randomized to receive a single, subcutaneous injection of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-6016a — DS-6016a will be administered as a single subcutaneous injection into the upper arm, upper part of the thigh, or abdominal wall
  Arms: DS-6016a dose level 1; DS-6016a dose level 2; DS-6016a dose level 3; DS-6016a dose level 4; DS-6016a dose level 5; DS-6016a dose level 6
Drug: Placebo — Placebo will be administered as a single subcutaneous injection into the upper arm, upper part of the thigh, or abdominal wall
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics of DS-6016a after subcutaneous injection in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects.
* Age ≥20 and ≤45 years upon providing informed consent.
* Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 at screening.

Exclusion Criteria:

* Have a history of hypersensitivity to any drugs or substances, or being idiosyncratic (eg, having penicillin allergy)
* Have alcohol or drug dependence, etc.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events | Day 1 through end of study, up to 8 weeks post-dose

SECONDARY OUTCOMES:
Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
Pharmacokinetic Parameter of Time to Reach Maximum Concentration (Tmax) of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
Pharmacokinetic Parameter of Area Under the Concentration-time Curve of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
  Area under the concentration-time curve from time 0 to last measurable time point (AUClast), time 0 to 336h (AUC336h), and time 0 to infinity (AUCinf) will be assessed.
Pharmacokinetic Parameter of Total Clearance (CL/F) of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
Pharmacokinetic Parameter of Terminal elimination half-life (t1/2) of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
Pharmacokinetic Parameter of Volume of Distribution (Vz/F) of Plasma DS-6016a Following Subcutaneous Administration of DS-6016a | Day 1 (pre-dose, 2 and 8 hours after the start of administration), Day 2 (24 and 36 hours after the start of administration), Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 12, Day 15, Day 18, Day 22, Day 29, Day 36, Day 43, Day 57
Proportion of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) | Day 1 (pre-dose), Day 29 and Day 57 post-dose
  The immunogenicity of DS-6016a will be assessed.
Proportion of Participants Who Have Treatment-emergent ADAs | Day 1 (pre-dose), Day 29 and Day 57 post-dose
  The immunogenicity of DS-6016a will be assessed.
Proportion of Participants Who Have Anti-host Cell Protein (HCP) Antibodies | Day 1 (pre-dose), Day 29 and Day 57 post-dose
  The immunogenicity of DS-6016a will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/